CLINICAL TRIAL: NCT03174353
Title: A Phase II Trial of Lanreotide for the Prevention of Postoperative Pancreatic Fistula
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Venu Pillarisetty, Professor of Surgery, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002777
Record Dates: First submitted 2017-05-26; First posted 2017-06-02 (Actual); Results first posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Leak; Pancreatic Fistula; Pancreaticoduodenal; Fistula; Pancreatectomy; Hyperglycemia
MeSH Terms: conditions — Pancreatic Fistula; Fistula; Hyperglycemia | interventions — lanreotide; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lanreotide arm (Experimental): Single arm study. A single deep subcutaneous dose of lanreotide (Somatuline Depot 120 Mg/0.5Ml) will be administered prior to planned resection on the day of surgery.
  Interventions: Drug: Lanreotide Prefilled Syringe

INTERVENTIONS:
Drug: Lanreotide Prefilled Syringe — All patients enrolled in this study will receive SOMATULINE DEPOT 120 mg immediately prior to planned pancreatic resection. The pharmacist will dispense loaded syringes of the study drug. The single preoperative dose will be given in the pre-surgical center at the University of Washington by a trained health care professional. The study drug will be injected via the deep subcutaneous route in the superior external quadrant of the buttock.
  Other Names: Somatuline Depot 120 Mg/0.5Ml Solution for Injection

SUMMARY:
This is a single arm investigator-initiated study designed to test the feasibility and potential efficacy of preoperative lanreotide to reduce the risk of postoperative abscess or pancreatic leak and fistula. All consenting patients undergoing planned elective pancreaticoduodenectomy or distal pancreatectomy for malignancy or suspected malignancy will be treated with a single deep subcutaneous dose of lanreotide prior to planned resection on the day of surgery. Following this intervention, care will be based on standard treatment protocols. Sixty-day mortality and morbidity will be collected for all patients.

DETAILED DESCRIPTION:
All patients enrolled in this study will receive SOMATULINE DEPOT 120 mg immediately prior to planned pancreatic resection. The pharmacist will dispense loaded syringes of the study drug. The single preoperative dose will be given in the pre-surgical center at the University of Washington by a trained health care professional. The study drug will be injected via the deep subcutaneous route in the superior external quadrant of the buttock.

Safety and efficacy will be assessed throughout the study period. Assessment for pancreatic and non-pancreatic complications will be made at the time of discharge and in follow-up by the attending surgeon. Patients will be evaluated in clinic postoperatively within 21 days of discharge for evaluation of the primary endpoint. The research team will perform long term follow-up by phone or in person with patients at 30 and 60 days (+/- 10 days at each time point).

SCREENING AND ENROLLMENT

Subjects undergoing planned elective pancreaticoduodenectomy or distal pancreatectomy for malignancy or suspected malignancy will be identified and screened for eligibility. Eligible patients who agree to participate will sign a written consent form at this time. At the initial visit, eligibility will be confirmed and documented in the study record. Informed consent will be obtained prior to enrollment utilizing the consent form.

STUDY PROCEDURES

1. Screening Visit (Day -60 to -1) Eligible patients will be identified at the Seattle Cancer Care Alliance (SCCA) and the University of Washington Medical Center (UWMC) surgical oncology clinics. At the screening visit, the Research Coordinator (RC) or one of the investigators will obtain signed informed consent. This will take place prior to any procedures being performed. Subjects will not receive any compensation for participation in the study. In addition, subjects will not incur any additional costs as a result of participation in the study.

   • Obtain and document consent from potential subject on study consent form

   • Review medical history to determine eligibility based on inclusion/exclusion criteria

   • Review medications history to determine eligibility based on inclusion/exclusion criteria

   • Perform physical examination: vital signs, weight, height

   • Collect, or obtain from routine care records, the following laboratory studies within 30 days prior to treatment:

   o Complete blood count with white blood cell differential and platelet counts;

   o Comprehensive profile; prothrombin time and activated partial thromboplastin time (PT&PTT)

   o Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to study drug administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
2. Preoperative Baseline (Day 0) The baseline visit will take place on the day of surgery, prior to the patient's operation and administration of the study drug. Some subjects initially consented into the study may be deemed ineligible on the day of surgery prior to drug administration. The study team will assess inclusion/exclusion criteria prior to drug administration.

   • Verify inclusion/exclusion criteria

   • Obtain demographic information, medical history/current condition, medication list

   • Collect serum pregnancy test for women of childbearing potential prior to drug administration, unless testing negative within prior 72 hours (for example, if testing was performed at Screening Visit within the previous 3 days), or testing has been performed for routine clinical care

   • Draw blood for correlative research (2 light green top tubes (10 ml)) prior to study drug administration (optional)
3. Preoperative Drug Administration (Day 0) The study drug will be administered and other study procedures performed after baseline procedures are conducted; prior to the surgery.

   • Administer the study drug
   * Administer Symptoms Questionnaire
   * Assess vital signs
   * Record results of pain on visual analog scale from chart
4. Intraoperative

   • Draw blood for correlative research (2 light green top tubes (10 ml)) intraoperatively immediately following resection (optional)
5. Postoperative Follow-up

5.a Hospital Stay (Postoperative Days 0-7) Subjects who receive the study drug but do not have a clinical resection performed during their surgery, will have no additional study procedures performed. The study team will review adverse events related to the study drug during the immediate postoperative hospital stay only.

Subjects who receive the study drug and have a clinical resection will be followed postoperatively for 60 days. The initial postoperative assessment will occur during the subject's hospital stay. Hospital stays will vary widely by patient, but are expected to range from 3-7 days. The study team will periodically review the patient chart for safety and outcomes as available for individual subjects during this timeframe.

* Record adverse events as reported by subject or observed by clinical team and/or investigator. See section 10.2 for list of information to be reviewed for adverse event monitoring
* Obtain medical history/current condition, medication list on the day of discharge
* Record results of physical examination on the day of discharge
* Collect the following laboratory studies, as available from routine care records:

  * Complete blood count with white blood cell differential and platelet counts;
  * Comprehensive profile; prothrombin time and activated partial thromboplastin time (PT&PTT)
* Assess vital signs
* Record results of pain on visual analog scale from chart
* Administer Symptoms Questionnaire on the day of discharge
* Record drain amylase levels from chart, as available
* Record drain output in ml from chart, as available
* Evaluate for day of drain removal from chart, as available

  5.b Clinic Follow-up Visit (Post discharge Days 1-21) Subjects will typically have a clinical follow-up appointment with their University of Washington (UW) Medicine surgical provider or an external provider within 1 - 21 days following discharge. There may be more than one clinical appointment during this timeframe. The study team will review patient charts and collect information on individual subjects as available from their clinical care. Subjects who are seen at UW Medicine will receive an in-person symptoms questionnaire to complete. Subjects who have their follow-up care performed external to UW Medicine will receive a phone call from the research coordinator (RC) between 1 and 21 after discharge to complete the symptoms questionnaire by phone. Records from external institutions will be obtained and reviewed for the time frame.
* Record adverse events as reported by subject or observed by clinical team and/or investigator
* Obtain medical history/current condition, medication list
* Record results of physical examination
* Collect from routine care records the following laboratory studies, as available:

  o Complete blood count with white blood cell differential and platelet counts;

  o Comprehensive profile; prothrombin time and activated partial thromboplastin time (PT&PTT)
* Assess vital signs
* Record results of pain on visual analog scale from chart
* Administer Symptoms Questionnaire

  6. Long Term Follow-up

  6.a Follow-up Phone Call (Postoperative Days 30 & 60) The RC will follow-up with all subjects by phone at approximately 30 and 60 days postoperative to identify missed complications. If the RC identifies a missed complication by phone, the investigator or co-investigator will then contact the subject with a second phone call to discuss the reported complications in more detail.

Patient charts will be reviewed throughout 60 days postoperative. Some subjects may receive their follow-up care outside of UW Medicine. In this case, records from external institutions will be obtained and reviewed for the timeframe.

* Record adverse events as reported by subject or observed by investigator.
* Obtain medical history/current condition, medication list
* Administer Symptoms Questionnaire
* Review clinical charts for complications, as available

SUBJECT WITHDRAWAL

Patients may voluntarily withdraw from the study or be dropped from it at the discretion of the investigator at any time. Patients may be withdrawn from the study if any of the following occur:

* Pregnancy discovered after enrollment, but prior to study drug treatment
* Protocol violation
* Subject withdrawal of consent
* Lost to follow-up
* Do not have clinical resection performed post drug administration
* Death

  1. Replacement of Subjects Subjects withdrawn from the study prior to administration of the study drug will be replaced. Subjects withdrawn from the study after administration of the study drug and who do not have a clinical resection performed will not be replaced. Other subjects withdrawn prior to complete 60-day follow up will not be replaced. If subjects do not respond to phone follow-up at 30 or 60 days, three repeated attempts will be made over the 10 days following each of these time points. Subjects who have incomplete follow up will be included with limited follow up.

BIOSTATISTICS

1. Sample Size and Power

   We estimate the final target sample size will be 98 patients. We aim to screen 154 patients and enroll n=123 patients into this single-arm study to test whether treatment with lanreotide reduces the risk of postoperative pancreatic fistula. Based upon a 20% probability of not proceeding with surgical resection after drug treatment due to findings of metastatic or unresectable disease at surgery, we anticipate that 123 treated patients will yield 98 evaluable patients.
2. Analysis Plan

As a primary method analysis, we will use a one-sample t-test to compare the rate of postoperative pancreatic fistula among the n=98 patients who were treated with lanreotide and underwent surgical resection against a published rate of 21% for patients treated with a placebo in another study, while 9% of patients treated with pasireotide experienced postoperative pancreatic fistula. The present study has 80% power (one-sided alpha = 0.05) to detect pancreatic fistula rates smaller than 11.5%, the approximate upper estimate of an 80% confidence interval of the pancreatic fistula rate of 9% in the study of pasireotide.

As a secondary exploratory analysis, we will use McNemar's test to compare the pancreatic fistula rate in the present study to that of historical controls at the same institution matched on pancreatic firmness and duct size.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age ≥ 18 years
* Candidate for planned elective pancreaticoduodenectomy or distal pancreatectomy for malignancy or suspected malignancy
* Able to provide informed consent
* Able to adhere to dose and schedule of visits
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to study drug administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects who are at risk of becoming pregnant must agree to use an effective method of contraception such as double barrier contraception, an injectable, combined oral contraceptive or an intra-uterine device (IUD). The subject must agree to use the contraception during the whole period of the study and for eight months after the last study drug administration. Non childbearing potential is defined as being postmenopausal for at least 1 year, or permanently sterilized at least 3 months before study entry.
* Male subjects must agree that, if their partner is at risk of becoming pregnant, they will use an effective method of contraception.

Exclusion Criteria:

* Use of disallowed concomitant medications
* Has been treated with a Somatostatin analogs (SSA) at any time prior to planned study drug administration, except if that treatment was for less than 15 days of short acting SSA or one dose of long acting SSA and the treatment was received more than 6 weeks prior to randomization
* Planned tumor enucleation or total pancreatectomy
* Pregnancy or breastfeeding
* Malabsorption syndrome, short bowel, or chologenic diarrhea uncontrolled by specific therapeutic interventions
* New York Heart Association (NYHA) Class III or IV congestive heart failure, unstable angina, sustained ventricular arrhythmia, advanced heart block, clinically significant bradycardia, or acute myocardial infarction within six months before enrollment
* Severe renal insufficiency as defined by a calculated creatinine clearance <30 mL/min
* Known allergic reactions to components of the study drug
* Has been treated with Peptide receptor radionuclide therapy (PRRT) at any time prior to randomization
* Treatment with systemic immunosuppressive medications, such as cyclosporine, tacrolimus, or prednisone (≥10 mg daily) within 3 months prior to dosing of study drug
* Treatment with another investigational drug within 10 days prior to dosing of study drug
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venu G Pillarisetty, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were recruited in the clinic, between February 2018 and February 2021.
Groups:
- Lanreotide Arm: Single arm study. A single deep subcutaneous dose of lanreotide (Somatuline Depot 120 Mg/0.5Ml) will be administered prior to planned resection on the day of surgery.
  Lanreotide Prefilled Syringe: All patients enrolled in this study will receive SOMATULINE DEPOT 120 mg immediately prior to planned pancreatic resection. The pharmacist will dispense loaded syringes of the study drug. The single preoperative dose will be given in the pre-operative area at the University of Washington by a trained health care professional. The study drug will be injected via the deep subcutaneous route in the superior external quadrant of the buttock.
Period: Overall Study
Arm/Group | Lanreotide Arm
Started | 114
Completed | 98
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Lanreotide Arm
Number analyzed (Participants) | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 96
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 85
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 98

OUTCOME MEASURES:

1. Primary Outcome: Combined Clinically Significant Postoperative Pancreatic Fistula and Intra-abdominal Abscess
Description: Reduction in the incidence of intraabdominal abscess or development of clinically significant (grade B or C) pancreatic fistula within 60 postoperative days. The grading of the primary outcome measure is based on a method published by the International Study Group of Pancreatic Surgery (ISGPS) in 2005 and then revised in 2016. As this study was developed prior to the revision, the 2005 version was used. This system for grading pancreatic fistula is based on progressively increasing severity of the complication from grade A to C. Grade Grade A fistula are characterized by elevated amylase detected within fluid coming from drain(s) placed at the time of surgery. Grade B fistula require change in patient management such as need for drain placement or institution of antimicrobial therapy, while grade C fistula are associated with severe clinical signs or symptoms such as sepsis. Please refer to page 12 of the study protocol for further details.
Time Frame: Measured throughout 60 days
Population: Patients undergoing pancreaticoduodencectomy or distal pancreatectomy for malignancy or suspected malignancy
Measure: Count of Participants; unit: Participants
Groups:
- Lanreotide Arm: Patients undergoing pancreaticoduodencectomy or distal pancreatectomy for malignancy or suspected malignancy
Arm/Group | Lanreotide Arm
Number analyzed (Participants) | 98
Participants | 8

2. Secondary Outcome: Biochemical Leak (Grade A Postoperative Pancreatic Fistula)
Description: Grade A pancreatic fistula will be defined based on principles noted in evaluation of Primary endpoint. Grade A fistula are characterized by elevated amylase detected within fluid coming from drain(s) placed at the time of surgery, but do not cause deviation from standard post-operative recovery.
Time Frame: Measured throughout 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lanreotide Arm
Number analyzed (Participants) | 98
Participants | 12

3. Secondary Outcome: Overall Postoperative Morbidity
Description: Overall morbidity was defined based on the National Surgical Quality Improvement Program (NSQIP) templates. This measure counts the number of participants who had a complication during the 60-day study period.
Time Frame: Measured throughout 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lanreotide Arm
Number analyzed (Participants) | 98
Participants | 26

ADVERSE EVENTS:
Time Frame: The adverse event were collected up to 60 days following operation.
Arm/Group | Lanreotide Arm
All-Cause Mortality (participants affected / at risk) | 0/98
Serious Adverse Events (participants affected / at risk) | 8/98
Other Adverse Events (participants affected / at risk) | 2/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Arm (N=98)
Clinically significant postoperative pancreatic fistula (Surgical and medical procedures) | 8 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Arm (N=98)
Drug-related adverse event (Skin and subcutaneous tissue disorders) | 2 (2) — Skin reaction

LIMITATIONS AND CAVEATS:
Single arm Single center Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03174353/Prot_SAP_001.pdf